CLINICAL TRIAL: NCT02044458
Title: A Randomized Control Trial of Foley Catheter Placement for Induction of Labor: Stylette Versus no Stylette
Brief Title: Foley Catheter for Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #13-46E :Foley Catheter
Record Dates: First submitted 2013-07-09; First posted 2014-01-24 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-03

CONDITIONS: Foley Catheterization; Induction of Labor; 5 French Stylette
Keywords: Foley Catheterization; Induction of Labor; 5 French Stylette

ARMS (2):
- Stylette (Active Comparator): Stylette: a thin wire inserted into a catheter to maintain rigidity, used to guide the insertion of the Foley catheter.
  Interventions: Device: Stylette
- No Stylette (No Intervention): No Stylette: 22 French Foley catheter placed without stylette or guide.

INTERVENTIONS:
Device: Stylette — use of stylette for successful insertion of foley catheter for induction of labor
  Other Names: 5 French stylette; Rigid catheter guide; Urethral manipulator (TVT procedure)
  Arms: Stylette

SUMMARY:
Study Design:

Allocation: 2 arms Intervention Model: Single Group Assignment Masking: Open Label Primary Purpose: Treatment

Detailed Description

The utilization of a Foley catheter for induction of labor is well established. There are two techniques readily used for placing a Foley catheter. The most common method is under direct visualization of the cervix during a sterile speculum examination and the other method is to place a catheter during a digital cervical examination.

Studies have reported the use of a rigid stylette (a thin wire inserted into a catheter to maintain rigidity) to guide the insertion of the Foley catheter decreases failure rate. The Foley catheter plus rigid stylette technique seems to be an efficient and safe method for labor induction. However, to our knowledge there is no study that assesses the difference between the standard digital placement of a Foley catheter versus the digital placement of a Foley catheter with stylette.

DETAILED DESCRIPTION:
Outcomes:

Primary Outcome Measures:

• The duration of insertion between the Foley catheter groups with and without a stylette.

Secondary Outcome Measures:

• Pain assessed by visual analogue scale (VAS), in women randomly allocated to rigid stylette or no rigid stylette placement of a Foley catheter for induction of labor.

Tertiary Outcome Measure:

• Compare the failure rate of the placement of a Foley catheter for induction of labor in women randomly allocated to rigid stylette or no rigid stylette

Design and Methods:

The decision to proceed with induction of labor with Foley catheter will be made by the attending obstetrician caring for the patient. Women requiring induction of labor will be consented to be in the study when the need for induction is confirmed. After obtaining informed consent, the nurse involved in the patient care will be notified of the patient's participation in the study. Random assignment to either a Foley bulb with 5 French stylette versus without will be achieved by the resident physician selecting the next sealed, opaque envelopes containing the assignment information. The envelopes only show the randomization number on the outside. Envelopes will be kept on the Labor and Delivery ward. It will be impossible for the performing physician or the patient to be blinded to the condition of the study due to the instruments needed for the different techniques. The performing physician will be decided prior to the envelop selection and will be the same resident physician who obtained the patient's Bishop Score. A 22 French Foley catheter will be used in both groups of the study. A 5 French stylette (also known as a rigid catheter guide or urethral manipulator used in the TVT procedure) will be used in the group assigned to the stylette.

Pre-induction cervical examination and assessment of Bishop score to be done by an OB/GYN resident physician (PGY 2-4) on the labor and delivery ward. Insertion technique for the Foley bulb with or without the 5 French stylette will be started in the same way. The patient will be placed in the dorsal lithotomy position. The labor bed will be disassembled in the normal fashion as is done for laboring patients with the foot of the bed removed. The patient's feet will then be placed in foot rests. The OB/GYN resident (PGY 2-4) will then perform a vaginal examination to identify the internal os. The Foley catheter, with or without stylette, will then be guided over the examiner's hand and into the endocervix. When the Foley balloon is past the internal os, the balloon will be inflated with 50cc normal saline. The Foley catheter will be placed on gentle traction and taped to the right medial thigh of the patient. Gentle traction will be reapplied every 30-60 minutes with reapplication of the tape to the right medial thigh by the Registered Nurse. This will be continued until expulsion of the Foley balloon or at a maximum duration of 12-24 hours. After expulsion of the Foley balloon, induction of labor will be further carried out with oxytocin infusion and/or with artificial rupture of membranes.. If the Foley catheter is removed at 24 hours status post insertion, the procedure will counted as a failed induction of labor with the Foley catheter and other methods of induction will be continued (i.e. Misoprostol, Artificial rupture or membranes, Oxytocin, etc.).

The time will begin at the start of the vaginal examination for placement of the Foley catheter and end after the balloon has been filled completely with saline.

Timeframe: Participants will be enrolled from April 2013 to January 2014 or until we have successfully enrolled 128 (64 per group) participants in the study. Data will be collected throughout the duration of the study to allow for all information from the hospital stay to be entered in the patient's medical record. Data analysis will occur from January 2014 to February 2014. Data presentation could occur up to 2 years after the complete of the study.

Data Collection:

The following variables will be recorded: Age; Race (0=NA; 1=Caucasian; 2=African American/Black; 3=Hispanic; 4=Asian 5=Other); BMI; Gravidity and Parity; Gestational Age; Reason for Indication for Induction (0=NA; 1=Post-term pregnancy; 2=Spontaneous Rupture of the Membranes; 3=Maternal disease; 4=Fetal indications; 5=Psychosocial parameters; 6= In vitro fertilization; 7=Advanced maternal age; 8 Maternal Request; 9=Other); History of Previous Cesarean Deliveries; Diabetes mellitus (0=NA; 1=Type I; 2=Type II; 3=Prediabetes; 4=GDM); Hypertensive disorders (0=NA; 1=Chronic HTN; 2= Gestational HTN; 3=Mild Preeclampsia; 4=Severe Preeclampsia; 5=Eclampsia); Renal Disease (0=No; 1=Yes); Other Comorbidities (0=No; 1=Yes); Documented Chorioamnionitis (0=No; 1=Yes); Epidural (0=No; 1=Yes); Inadvertent Rupture of Membranes (0=No; 1=Yes); Type of Delivery; Pain Assessment (0-10); Patient Satisfaction; Type of Delivery.

Points of time recorded will be: Time of insertion (Placement of Foley catheter); Time of expulsion of catheter; Time taken to place catheter; Time oxytocin started; Time oxytocin ended; Duration of treatment (Insertion to expulsion); Duration of induction (induction to delivery); Duration of oxytocin.

All variables will be recorded on an Excel spreadsheet by the resident physician or study coordinator. See attached example.

ELIGIBILITY:
Inclusion Criteria:

* Singleton fetus
* Cephalic presentation
* Indicated or Post-Estimated Date of Confinement
* Induction of labor with a Bishop score < 5

Exclusion Criteria:

* Low lying placenta
* Undiagnosed vaginal bleeding
* History of induction or pre-induction agent during the same pregnancy
* Signs or symptoms of infection (i.e. Maternal fever)
* Rupture of membranes
* Multiple gestation
* Women with an urgent or emergent clinical situation in which the medical staff caring for the patient determines that obtaining consent would interfere with the patient's clinical care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danish S Siddiqui, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Sinia Medical Center, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stylette | No Stylette
Started | 65 | 69
Completed | 62 | 61
Not Completed | 3 | 8
Not completed — Protocol Violation | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stylette | No Stylette | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (5.56) | 26.9 (6.98) | 26.9 (6.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 123
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic | 15 | 8 | 23
  African-American non-Hispanic | 38 | 41 | 79
  Hispanic/Latina | 6 | 10 | 16
  Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 62 | 61 | 123

OUTCOME MEASURES:

1. Primary Outcome: Duration of Insertion Between Foley Catheter Groups With and Without a Stylette.
Description: Difference in insertion times between women randomly allocated to ridged stylette or no ridged stylette. Patient's may have experienced multiple insertions only if a patient failed initial randomized insertion method. Subsequent treatment methods were used when a patient failed and time was summarized as length of time of attempt. Failure was defined as either inadvertent amniotomy, excessive time in placement (subjectively determined by the provider using the catheter), or excessive patient pain (subjectively defined by the provider but based on patient response).
Time Frame: Followed throughout patient's hospital stay, approximately 10 days
Population: The insertion time of two failed attempts with no stylette were not recorded.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Stylette | No Stylette
Number analyzed (Participants) | 62 | 59
minutes
  Successful insertion attempts | 1.72 [1.25 to 3.30] | 1.88 [1.33 to 3.12]
  Failed insertion attempts | 6.55 [3.80 to 11.6] | 5.00 [3.00 to 7.18]
Statistical Analysis 1: Comparison: Stylette; Test type: Superiority or Other; p = .70, t-test, 2 sided

2. Secondary Outcome: Pain Assessed by Visual Analog Scale (VAS)
Description: To compare the pain assessed by visual analogue scale(VAS), in women randomly allocated to ridged stylette or no ridged stylette. Patient-assessed pain level was determined by verbally asking patients to assess their pain (on a scale from 0-10 [no pain-worst pain]) following taping of the catheter tail. Pain was only assessed once.
Time Frame: Followed throughout patient's hospital stay, approximately 10 days
Population: The pain level of one successful attempt with stylette was not recorded.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Stylette | No Stylette
Number analyzed (Participants) | 61 | 61
units on a scale | 4.90 [4.22 to 5.58] | 4.43 [3.59 to 5.27]
Statistical Analysis 1: Comparison: Stylette; Test type: Superiority or Other; p = .38, t-test, 2 sided

3. Other Pre Specified Outcome: Failure Rates of the Placement of a Foley Catheter
Description: To compare the failure rate of the placement of a Foley catheter for the induction of labor in women randomly allocated to rigid stylette or no stylette
Time Frame: Followed throughout patient's hospital stay, approximately 10 days
Measure: Number; unit: failed attempt
Arm/Group | Stylette | No Stylette
Number analyzed (Participants) | 62 | 61
failed attempt | 7 | 9
Statistical Analysis 1: Comparison: Stylette; Test type: Superiority or Other; p = .57, Chi-squared

ADVERSE EVENTS:
Time Frame: Study Duration; June 2013-December 2014 (1 year, 6 months)
Description: Serious and other adverse events were collected and assessed, but none were observed.
Arm/Group | Stylette | No Stylette
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/69
Other Adverse Events (participants affected / at risk) | 0/65 | 0/69

LIMITATIONS AND CAVEATS:
Did not enroll enough subjects to achieve sufficient power for every test performed or to study outcomes with low event rates. Insertion time and failure may be influenced by providers comfort with insertion technique. Women were from a single site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No